CLINICAL TRIAL: NCT00748501
Title: A Phase 2 Repeat-Dosing Clinical Trial of SB-509 in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Clinical Trial of SB-509 in Subjects With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB-509-0801
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis,; ALS,; Lou Gehrig's Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Active Comparator): SB-509 drug administration via IM injection of neck, arms, and legs
  Interventions: Drug: SB-509
- Cohort 2 (Active Comparator): SB-509 drug administration via IM injection of legs
  Interventions: Drug: SB-509

INTERVENTIONS:
Drug: SB-509 — Intramuscular injection of 60 mg of SB-509. Two doses on Day 0 and Day 90.

SUMMARY:
The purpose of the study is to evaluate the effects of the investigational drug, SB-509 on progression of the disease in subjects with ALS

DETAILED DESCRIPTION:
SB-509 contains the gene (DNA-a kind of biological "blueprint") for a protein. When a study doctor injects SB-509 into the muscles of your neck, arms and/or legs, the drug enters the muscle and nerve cells around the injection sites and causes these cells to make a protein. This protein causes your cells to increase production of one of your own protein called vascular endothelial growth factor(VEGF-A), which may improve the structure and function of nerves and muscles. In addition, there are changes in the levels of 28 additional proteins in your cells. These proteins function to promote the growth of cells, are structures in cells, help synthesize products, and affect immune cells, and some have unknown functions. This increase in your own VEGF proteins may protect and repair the damaged nerves and muscles caused by ALS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18 and 85 with clinical diagnosis of ALS
* Forced Vital Capacity (FVC) > 60% of predicted
* Less than 3 years of ALS since the onset of the first symptom with clinical evidence of limb muscle atrophy and weakness.
* Subjects taking Riluzole must have been at a stable dose for at least 30 days with no evidence of toxicity
* Female of childbearing potential and male of child-creating potential must agree to use a medically acceptable physical barrier (condom, diaphragm, and cervical cap) through the treatment phase and for at least 30 days after the last study treatment.

Exclusion Criteria:

* Women who are pregnant or currently breast-feeding
* Dependent upon invasive or non-invasive artificial ventilation
* Patients with bulbar onset ALS or with other active neuromuscular/ neurodegenerative diseases.
* Type 1 or Type 2 diabetes.
* Evidence of chronic or active heart, liver, kidney, or lung diseases, or Age-related macular degeneration.
* Current or history of known immune or immunodeficiency disorders
* Patients with cognitive impairment with significant decision making incapacity, or major depression, or schizophrenia, or dementia (e.g. Alzheimer's disease).
* Malignancy or history of malignancy, except it has been in complete remission for at least 5 years
* Pre-cancerous conditions (e.g. Barrett's Esophagus, dysplasias) or benign tumors which have the potential for significant growth due to VEGF stimulation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of SB-509 on progression of the disease in subjects with ALS, as measured by the ALS Functional Rating Scale -Revised (ALSFRS-R). | 11 months

SECONDARY OUTCOMES:
To evaluate a) the effect of SB-509 on Forced Vital Capacity, Neurophysiologic Index, Manual Muscle Test, and survival. b) safety and tolerability of SB-509 in ALS. c) stem cell mobilization in subjects with ALS receiving SB-509. | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Ely Benaim, M.D., Study Director — Sangamo Therapeutics
Locations (6):
- United States (6):
  - Coordinated Clinical Research, La Jolla, California
  - University of California, Irvine; MDA ALS and Neuromuscular Center,, Orange, California
  - California Pacific Medical Center (CPMC), The Forbes Norris MDA/ALS Research Center, San Francisco, California
  - The University of Kansas Medical Center (KU), Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Nerve and Muscle Center of Texas, Houston, Texas